CLINICAL TRIAL: NCT05007782
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Denikitug (GS-1811), an Afucosylated Anti-CCR8 Monoclonal Antibody, as Monotherapy and in Combination With an Anti-PD-1 Monoclonal Antibody in Adults With Advanced Solid Tumors
Brief Title: Study of Denikitug (GS-1811) Given Alone or With Zimberelimab in Adults With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-570-6015; 2022-501684-40 (Other: European Medicines Agency)
Record Dates: First submitted 2021-08-11; First posted 2021-08-16 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A - Denikitug Dose Escalation (Experimental)
  Interventions: Drug: Denikitug
- Part B - Mandatory Paired Tumor Biopsy (Experimental)
  Interventions: Drug: Denikitug
- Part C: Denikitug + Zimberelimab Dose Escalation (Experimental)
  Interventions: Drug: Denikitug; Drug: Zimberelimab
- Part D: Denikitug + Zimberelimab Dose Expansion (Experimental)
  Interventions: Drug: Denikitug; Drug: Zimberelimab
- Part E: Denikitug Monotherapy Dose Expansion (Experimental)
  Interventions: Drug: Denikitug
- Part F: Denikitug Monotherapy and In Combination With Zimberelimab In Select Dose and Schedule (Experimental)
  Interventions: Drug: Denikitug; Drug: Zimberelimab

INTERVENTIONS:
Drug: Denikitug — Administered Intravenously
  Other Names: GS-1811
Drug: Zimberelimab — Administered Intravenously
  Arms: Part C: Denikitug + Zimberelimab Dose Escalation; Part D: Denikitug + Zimberelimab Dose Expansion; Part F: Denikitug Monotherapy and In Combination With Zimberelimab In Select Dose and Schedule

SUMMARY:
This is a first-in-human (FIH) study to evaluate the safety and tolerability and to determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of denikitug (also known as GS-1811) as monotherapy and in combination with zimberelimab in participants with advanced solid tumors.

This study will be conducted in 6 parts (Parts A, B, and E: monotherapy, Parts C and D: combination therapy, and Part F for both monotherapy and combination therapy) in participants with advanced solid tumors who have received, been intolerant to, or been ineligible for all treatments known to confer clinical benefit or in participants with select solid tumors.

DETAILED DESCRIPTION:
Part D allocation for 1 cohort will be randomized.

ELIGIBILITY:
Key Inclusion Criteria:

* Disease:

  * Part A: Individuals with histologically or cytologically confirmed advanced solid tumors who have received, been intolerant to, or been ineligible for all treatment known to confer clinical benefit.
  * Part B: Individuals with histologically or cytologically confirmed select indications who have received, been intolerant to, or been ineligible for all treatment known to confer clinical benefit.
  * Part C: Individuals with histologically or cytologically confirmed advanced solid tumors who have received, been intolerant to, or been ineligible for all treatments known to confer clinical benefit or whose disease is indicated for anti- programmed cell death protein 1 or programmed cell death ligand 1 (PD-[L]1) monoclonal antibody monotherapy.
  * Part D: Individuals with pathologically confirmed select advanced solid tumors.
  * Part E: Individuals with pathologically confirmed select advanced solid tumors. Participants must have received, have been intolerant to, or have been ineligible for all treatment known to confer clinical benefit.
  * Part F: Individuals with pathologically-confirmed select advanced solid tumors. Participants must have received, have been intolerant to, or have been ineligible for all treatments known to confer clinical benefit; or, for participants who will undergo combination therapy, have disease which is indicated for anti-PD-(L)1 mAb monotherapy.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 for individuals in Parts A, B, and C, and 0 or 1 for individuals in Parts D, E, and F.
* Adequate organ function.
* Male individuals and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use methods of contraception.
* Tissue requirement:

  * Parts A, C, D, E and F: Must provide pre-treatment adequate tumor tissue sample prior to enrollment.
  * Part B and select participants in Parts C and F: Must have fresh pre-treatment and on-treatment biopsies for biomarker analysis.

Key Exclusion Criteria:

* Concurrent anticancer treatment.
* Any anti-cancer therapy, whether investigational or approved, within protocol specified time prior to initiation of study including: immunotherapy or biologic therapy (< 28 days), chemotherapy (< 21 days), targeted small molecule therapy (< 14 days), hormonal therapy or other adjunctive therapy (< 14 days) or radiotherapy (< 21 days).
* Any prior CCR8 directed therapy.
* Prior allogeneic tissue/solid organ transplantation, including allogeneic stem cell transplantation. Exception: prior corneal transplant without requirement for systemic immunosuppressive agents is allowed.
* Concurrent active malignancy other than nonmelanoma skin cancer, curatively resected carcinoma in situ, localized prostate cancer, or superficial bladder cancer after undergoing potentially curative therapy with no evidence of disease. Individuals with other previous malignancies are eligible if disease-free for > 2 years.
* History of intolerance, hypersensitivity, or treatment discontinuation due to severe immune-related adverse events (irAEs) on prior immunotherapy.
* History of autoimmune disease or active autoimmune disease requiring systemic treatment within 2 years.
* History of pneumonitis, interstitial lung disease, or severe radiation pneumonitis (excluding localized radiation pneumonitis).
* Active and clinically relevant bacterial, fungal, or viral infection that is not controlled or requires IV antibiotics.
* Active hepatitis B virus (HBV) and/or hepatitis C virus (HCV), and/or human immunodeficiency virus (HIV).
* Positive serum pregnancy test or breastfeeding female.
* Live vaccines within 30 days prior to first dose.
* Significant cardiovascular disease.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs) in Part A and C | Day 1 Through Day 21
Percentage of Participants Experiencing Adverse Events (AEs) According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | First dose to End of Treatment (up to 12 months for monotherapy and 24 months for combination therapy) plus 90 days
Percentage of Participants Experiencing Laboratory Abnormalities According to the NCI CTCAE v5.0 | First dose to End of Treatment (up to 12 months for monotherapy and 24 months for combination therapy) plus 90 days

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax) for Denikitug | Day 1 Up to End of Treatment (up to 12 months for monotherapy and 24 months for combination therapy) plus 90 days
PK Parameter: Minimum Observed Concentration (Cmin) for Denikitug | Day 1 Up to End of Treatment (up to 12 months for monotherapy and 24 months for combination therapy) plus 90 days
PK Parameter: Time of Maximum Observed Concentration (Tmax) for Denikitug | Day 1 Up to End of Treatment (up to 12 months for monotherapy and 24 months for combination therapy) plus 90 days
PK Parameter: Area Under the Concentration-time Curve (AUC) for Denikitug | Day 1 Up to End of Treatment (up to 12 months for monotherapy and 24 months for combination therapy) plus 90 days
Percentage of Participants who Developed Antidrug Antibody (ADA) Against Denikitug | Day 1 Up to End of Treatment (up to 12 months for monotherapy and 24 months for combination therapy) plus 90 days
Objective response rate (ORR) in Part D | Day 1 Up to End of Treatment (24 months)
  Objective response rate is defined as the proportion of participants who achieve complete response (CR) or partial response (PR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Disease control rate (DCR) | Day 1 Up to End of Treatment (24 months)
  Disease control rate is defined as the proportion of participants who achieve CR, PR, or stable disease (SD) as assessed by RECIST Version 1.1
Time to response (TTR) | Day 1 Up to End of Treatment (24 months)
  Time to response is defined as the time from the first dose of Denikitug in combination with Zimberelimab to the first documentation of CR or PR that is subsequently confirmed
Duration of response (DOR) | Day 1 Up to End of Treatment (24 months)
  Duration of response is defined as the time from the first documentation of CR or PR to the earlier of the first documentation of definitive progressive disease (PD) or death from any cause, if applicable.
Progression-free survival (PFS) | Day 1 Up to End of Treatment (24 months)
  Progression-free survival is defined as the time from the first dose of Denikitug in combination with Zimberelimab to the earlier of the first documentation of definitive PD or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (26):
- United States (10):
  - University of California San Diego, La Jolla, California
  - Stanford Cancer Center, Palo Alto, California
  - Smilow Cancer Center, New Haven, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Sarah Cannon Research Institute at Mary Crowley, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - University of Wisconsin Clinical Sciences Center, Madison, Wisconsin
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- University Health Network, Princess Margaret Cancer Centre, Toronto, Canada
- Spain (5):
  - Hospital Universitari Vall d´Hebrón, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Clinica Universidad de Navarra, Pamplona
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Chi Mei Hospital, Liouying, Tainan
  - National Taiwan University Cancer Center (NTUCC), Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Tzu Chi General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-570-6015